CLINICAL TRIAL: NCT04875910
Title: Could Telerehabilitation be a Promising Tool in Improving Walking and Balance Among Stroke Survivors? "Case Study"
Brief Title: Effectiveness of Telerehabilitation in Improving Walking and Balance Among Stroke Survivors?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Emtenan Alsadhan, Master's student, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tele-rehabilitaion exercises
Record Dates: First submitted 2021-05-01; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke survivors participants (Experimental): Subjects who have been diagnosed with stroke 6 months or more.
  1)Either right and left hemiparesis. 2) Subjects able to walk with or without assistive device. 3) age between 40-80. 4) Subjects can understand and follow commands.
  Exclusion criteria is: 1) subjects with uncontrolled Blood pressure, heart rate or breathing problems. 2) Having an orthopedic problem or
  Interventions: Other: Home-based exercise program

INTERVENTIONS:
Other: Home-based exercise program — The exercise program will include task specific training to improve balance and the training will progress every two weeks. A Physical therapist will be following up and monitoring the participants adherence to the training by audio or video call.
  The exercise program for Week 1: Sit to Stand 5 times, Steps forward, backward and to the sides 5 times, 10 meters walk. 45 minutes session /3 times per week. Week 2: Sit to stand 10 times, Steps forward, backward and to the sides 5 times , Sit and reach 5 min for each hand and walk for 15 meters. 45 minutes session, 3 times per week. Week3 Sit to stand 10 times, Step on bench 5 times, Stand and reach 5 and walk for 15 meters. 45 minutes session, 3 times per week. Week 4 Stand and reach 5 times, Step on bench 10 times, climbing stairs (5 steps flight stairs up and down) and walk for 20 meters. 50 minutes session, 3 times per week.

SUMMARY:
A good rehabilitation program may not be accessible for all individuals living with stroke due to cost, transportation and compliance. Telerehabilitation is an alternative health care program that may help in overcoming this issue. In this study we aim to find if the use of telerehabilitation in Saudi Arabia would improve balance and walking in stroke survivors during this pandemic.

DETAILED DESCRIPTION:
Background: Rehabilitation program is commonly provided after stroke to improve functional outcomes. A good rehabilitation program may not be accessible for all individuals living with stroke due to cost, transportation and compliance. Telerehabilitation is an alternative health care program that has been used to provide therapy for stroke survivors living in rural areas. With COVID-19 pandemic, many stroke survivors have lost their access to rehabilitation. Therefore, telerehabilitation may help in overcoming this issue. In this study we aim to find if the use of telerehabilitation in Saudi Arabia would improve balance and walking in stroke survivors during this pandemic.

Methods: 2 stroke survivors ( male and female/ >6 months post stroke) are included in this case study. Participants will receive a task-specific activity training (3days/week moderate exercises for 4 weeks) Both participants will provide feedback through questionnaires pre and post the 4 weeks intervention. We will use the Activities- specific balance confidence (ABC) scale, Lower limb functional scale (LEFS) and Stroke severity quality of life scale ( SS-Qol).

• Intervention: The participants will follow a home-based exercise through videos with follow up from the therapists for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been diagnosed with stroke 6 months or more.
* Either right or left hemiparesis.
* Subjects able to walk with or without assistive device.
* age between 40-70. 5) Subjects can understand and follow commands.

Exclusion Criteria:

* subjects with uncontrolled Blood pressure, heart rate or breathing problems.
* Having an orthopedic problem or pain that limits walking and standing.
* Subject with vestibular disorders.
* Subjects with cognitive disorders. 5) Subjects with hemi spatial neglect

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Change of balance confidence -The Activities- specific balance confidence (ABC) scale | pre and post intervention (1st and 4th week)
  Consists of 16 items scored from 0% to 100%, with 0 % equate no confidence and 100% equate total confidence. The higher score indicates higher balance confidence

SECONDARY OUTCOMES:
Change in lower extremity function - The lower extremity functional scale (LEFS) | pre and post intervention (1st and 4th week)
  consisted of 20 question to evaluate the lower limb functional impairment.The lower score equates greater disability
Change in Quality of life - Stroke Specific Quality Of Life scale (SS-QOL | pre and post intervention (1st and 4th week)
  measure aspects related to quality of life and designed specifically for stroke survivors

CONTACTS AND LOCATIONS:
Overall Officials: Almarwani, PhD, Study Director — Assistant professor at King Saud university
Locations (1):
- King Saud university, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided